CLINICAL TRIAL: NCT05358756
Title: A Phase 1, Open-label, Randomized, 3-period, 3-sequence, Single-dose Crossover Bioavailability and Food Effect Study of SACT-1 (Rilpivirine Suspension) and Edurant® Tablets in Healthy Adult Volunteers
Brief Title: A Study of Bioavailability and Food Effect of SACT-1 and Edurant® Tablets in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptorum International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12190001
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Rilpivirine; Tablets

STUDY DESIGN:
Intervention Model Description: Each of the following treatments were given to subjects in a randomized sequence:
  Treatment A: SACT-1, 150 mg rilpivirine oral suspension (30.0 mg of rilpivirine [equivalent to 33.0 mg of rilpivirine hydrochloride] in each mL), fasted Treatment B: SACT-1, 150 mg rilpivirine oral suspension (30.0 mg of rilpivirine [equivalent to 33.0 mg of rilpivirine hydrochloride] in each mL), fed Treatment C: Edurant, 150 mg (6 × 25 mg rilpivirine, oral tablets), fed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A :Fasted (Experimental): A single adminstration of SACT-1 (150 mg rilpivirine oral suspension) after a supervised overnight fast of at least 10 hours.
  Interventions: Drug: SACT-1
- Treatment B: Fed (Experimental): A single adminstration of SACT-1 (150 mg rilpivirine oral suspension) after a supervised overnight fast of at least 10 hours followed by a high-fat, high calorie meal (fed).Subjects started the standardized high-fat, high-calorie breakfast 30 minutes prior to dosing and consumed this meal within the 30 minutes before dosing.
  Interventions: Drug: SACT-1
- Treatment C: Fed (Active Comparator): Adminstartion of Edurant, 150 mg (6 × 25 mg rilpivirine, oral tablets), after a supervised overnight fast of at least 10 hours followed by a high-fat, high calorie meal (fed).Subjects started the standardized high-fat, high-calorie breakfast 30 minutes prior to dosing and consumed this meal within the 30 minutes before dosing.
  Interventions: Drug: EDURANT 25Mg Tablet

INTERVENTIONS:
Drug: SACT-1 — Single administartion of 150mg SACT-1
  Arms: Treatment A :Fasted; Treatment B: Fed
Drug: EDURANT 25Mg Tablet — Single administartion of six EDURANT 25mg tablets (Total 150mg)
  Arms: Treatment C: Fed

SUMMARY:
This was a Phase 1, open-label, randomized, single center, 3-period, 3-sequence, single-dose crossover bioavailability and food effect study between SACT-1 and Edurant® tablet.

DETAILED DESCRIPTION:
The subject population included 16 healthy subjects (11 male, 5 female) who received each of the following treatments in a randomized sequence:

Treatment A: SACT-1, 150 mg rilpivirine oral suspension (30.0 mg of rilpivirine [equivalent to 33.0 mg of rilpivirine hydrochloride] in each mL), fasted Treatment B: SACT-1, 150 mg rilpivirine oral suspension (30.0 mg of rilpivirine [equivalent to 33.0 mg of rilpivirine hydrochloride] in each mL), fed Treatment C: Edurant, 150 mg (6 × 25 mg rilpivirine, oral tablets), fed

On the morning of Day 1 of each study period, subjects received a dose of either Treatment A, Treatment B, or Treatment C after a supervised overnight fast of at least 10 hours (fasted) or after a supervised overnight fast of at least 10 hours followed by a high-fat, high calorie meal (fed). In the fed arms of the study, subjects started the standardized high-fat, high-calorie breakfast 30 minutes prior to dosing and consumed this meal within the 30 minutes before dosing.

Blood samples were collected at pre-dose and at specified time points over 240 hours after dosing in each study period. Subjects were confined at the clinical facility from check-in until after the 48-hour blood sample collection and returned to the clinic for the 96-, 168- and 240-hour blood samples in each study period. The interval between doses was 14 days.

The plasma concentrations of rilpivirine were measured by the bioanalytical facility using a fully validated analytical procedure. Statistical analysis using an average bioavailability approach was performed to estimate the bioavailability of the test formulation relative to the reference product under fed conditions. The bioavailability of the test product under fasted and fed conditions was also compared.

For evaluation of the safety endpoint, the following assessments were performed throughout the study: collection of medication history and Adverse Events (AEs), laboratory tests (including pregnancy testing), vital signs, physical examination, and 12-lead electrocardiograms (ECGs). PK-ECG correlation analysis was performed to evaluate the correlation between drug concentrations and time-matched baseline corrected values for QTc interval, ΔQTcF and ΔQTcB.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers ≥ 18 years of age.
2. Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation or hysterectomy), or who agree to use effective contraceptive methods throughout the course of the study and for 30 days after the last dose of study drug. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea and a serum FSH concentration ≥ 40 IU/L), or at least 6 weeks following surgical menopause (bilateral oophorectomy).
3. Females of childbearing potential and male subjects with female partners of childbearing potential must agree to use at least 1 of the following acceptable birth control methods during the study and for at least 30 days after the last dose:

   1. IUD in place for at least 3 months.
   2. Abstinence (not having heterosexual vaginal intercourse).
   3. Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening and through study completion and for 30 days after the last dose of study drug.
   4. Stable hormonal contraceptive for at least 3 months prior to study and through study completion (an additional barrier method must be used during the study) and for 30 days after the last dose of study drug. Oral contraceptive use is not permitted in this study.
   5. Monogamous relationship with a vasectomized partner.
4. Able to understand and provide signed informed consent.
5. Normally active and otherwise judged to be in good health on the basis of medical history and physical examination.
6. Females of childbearing potential must have a negative serum hCG pregnancy test at screening.
7. BMI ≥ 19.0 and < 32.0.
8. Willing and able to consume the entire assigned meals, which include meat, dairy and carbohydrate components, within the designated time frames.
9. Subjects must have normal hepatic function at the Screening Visit, defined as the following:

   1. Alanine aminotransferase <1.5 × upper limit of normal (ULN); or
   2. Aspartate aminotransferase < 1.5 × ULN; and
   3. Total bilirubin level <1.5 × ULN.
10. Subjects must have creatinine within normal limits or, for subjects with levels above the laboratory normal value, the calculated corrected creatinine clearance must be ≥60 mL/min/1.73 m2 using the Cockcroft-Gault formula corrected for the body surface area.

Exclusion Criteria:

1. Known or suspected pregnancy, planned pregnancy, or lactation.
2. History of allergic reaction to rilpivirine or other related drugs.
3. Clinically significant illness or surgery within 4 weeks prior to dosing (including flu, flulike symptoms, diarrhea, vomiting).
4. Positive test for hepatitis B, hepatitis C, or HIV at screening
5. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
6. Any clinically significant abnormal laboratory test results found during medical screening.
7. A history of major mental illness that in the opinion of the Investigator may affect the ability of the subject to participate in the study.
8. Clinically significant history or presence of any gastrointestinal pathology (eg, chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (eg, diarrhea vomiting), liver or kidney disease, gastric bypass, gastric stapling, use of Lapband, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
9. Any history of or active neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease that is considered clinically significant by the Investigator.
10. Use of prescription medication within 14 days prior to administration of study drug or OTC medicines (including natural food supplements and vitamins) within 14 days prior to administration of study drug.
11. Use of any tobacco- or nicotine- containing product in the 3 months preceding the Period 1 dose administration.
12. Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
13. Recent history of (within the past 12 months), or strong potential for, alcoholic substance abuse. Alcohol abused will be defined as > 14 drinks per week (1 drink = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
14. Exposure to any investigational agent within 30 days prior to study entry.
15. Subjects who donated (standard donation amount or more) blood or blood products (with the exception of plasma as noted below) within 56 days prior to the study.
16. Subjects who have made a plasma donation with 7 days prior to the study.
17. Subject who has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.
18. Positive SARS-CoV-2 test.
19. Subject currently taking oral contraceptives (for contraceptive and/or other medical purposes).
20. Unable or unwilling, due to allergy, food intolerance, dietary preference, or dietary restriction, to eat the assigned meals.
21. Known diagnosis of a mood disorder.
22. Subject has received any vaccine within 14 days prior to administration of study drug, or has any vaccination scheduled during the study period (from screening up until scheduled end-of-study-visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability of SACT-1 and Edurant Tablet | Up to 240 hours after dosing in each study period
  Compare the relative bioavailability of 150 mg SACT-1 (oral suspension) under fasted and fed conditions to 150 mg Edurant® (6 × 25 mg rilpivirine, oral tablets) under fed conditions.

SECONDARY OUTCOMES:
Number of subjects with Adverse Events | Up to 14 days after the final dose of the study drug.
  Adverse event or AE means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) can be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. An AE can arise from any use of the drug (eg, off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.
The effect of food (fasted or fed condition) on potential QT prolongation from administration of a single dose of 150 mg rilpivirine in healthy adult subjects. | Up to 24 hours after dosing in each study period
  Pharmacokinetic - Electrocardiogram (PK-ECG) correlation analysis was performed to evaluate the correlation between drug concentrations and time-matched baseline corrected values for corrected QT (QTc) interval, ΔQTcF and ΔQTcB.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lee, PhD, Principal Investigator — Aptorum International Limited
Locations (1):
- Novum Pharmaceutical Research Services, Fargo, North Dakota, United States